CLINICAL TRIAL: NCT04156555
Title: Antibiotic-associated Gastrointestinal Side Effects and the Role of the Gut Microbiome
Brief Title: Antibiotic-Associated Diarrhea and the Role of Microorganisms in the Gut
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AAD-MB-01; AM/CT003/2018 (SRDUKAMR18C3) (Other Grant/Funding Number: Singhealth DukeNUS Academic Medical)
Record Dates: First submitted 2019-10-28; First posted 2019-11-07 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Antibiotic-associated Diarrhea
Keywords: amoxicillin-clavulanate; diarrhea; Gut microbiome
MeSH Terms: conditions — Diarrhea | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study drug (Experimental)
  Interventions: Drug: Amoxicillin-Clavulanate 875 Mg-125 Mg Oral Tablet

INTERVENTIONS:
Drug: Amoxicillin-Clavulanate 875 Mg-125 Mg Oral Tablet — Oral amoxicillin-clavulanate 1 g twice a day for total of 6 doses
  Other Names: Augmentin; Moxiclav

SUMMARY:
Amoxicillin-clavulanate is an antibiotic commonly prescribed to treat a myriad of community-acquired infections. One of the most common adverse effects of amoxicillin-clavulanate is antibiotic-associated diarrhea (AAD). Studies have shown that administration of antibiotics can cause disruption and changes in the diversity of microorganisms within the gut (gut microbiome), with overgrowth of "harmful" bacteria as a possible driver for AAD. How antibiotics specifically affect the gut microbiome to cause AAD in humans, however, remains unknown. The overall goal of the study is to characterize the changes in the gut microbiome over time, in subjects who develop AAD after antibiotic ingestion, and to further demonstrate that resolution of AAD is due to return of "friendly, anti-diarrhea bacteria". The study investigators will also measure the proteins produced by the gut bacteria, as a potential tool to help predict which individuals are at risk of AAD.

The investigators plan to recruit 30 healthy adult volunteers who will receive 3 days of oral amoxicillin-clavulanate, a very commonly prescribed antibiotic. Stool and blood samples will be collected throughout the study up to 28 days after antibiotic administration. The study investigators will measure and compare the changes in the gut microbiome and metabolic responses in order to identify the relationship between these changes and the onset of AAD. The results from this study will not only yield important scientific knowledge about the pathogenesis of AAD, but will also provide new leads to understand the interplay between the gut microbiome, immune-metabolism and AAD. These findings also have the potential to identify clinically important biomarkers to allow pre-identification of individuals at risk of AAD. If successful, this study could pave the way for personalized medicine for management of bacterial infections. This will help to prevent premature stoppage of antibiotic therapy due to diarrhea side effects, and reduce the risk of bacterial resistance from suboptimal treatment.

DETAILED DESCRIPTION:
All eligible subjects will proceed to Day 0, where they will receive study drug amoxicillin-clavulanate 1g twice a day for 3 days. Prior to administration of study drug on Day 0, stool sample and blood will be collected for microbiome and metabolomics & gene expression analysis respectively. Urine pregnancy test (for females subjects of child-bearing potential) will be performed prior to study drug administration. Baseline physical examination and vital signs will be done as well.

Subsequently, stool and blood samples will be collected on day 1, day 2, day 3, day 7, day 14, and day 28. Physical examination, vital signs, and review of adverse events will be done at each of the visits as well.

Volunteers will be monitored for symptoms of AAD throughout this period. All study subjects will be asked to keep a standardised patient diary up to day 28 or until symptom resolution whichever is longer. All other potential AEs will also be solicited for throughout study period. Subjects who develop AAD will be graded according to CTCAE version 5.0 criteria for AEs. The study drug Augmentin will be discontinued in subjects who develop AAD, defined as a passage of loose or watery stool at least 3 times in a 24-hour period. Management of AAD is at the discretion of the study team PI and co-Is, guided by severity and clinical indication for intervention. All medication prescribed for the management of AAD or other AEs will be documented in the medication/concomitant medication clinical record form.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults, 21-40 years of age at time of screening
2. Satisfactory baseline medical assessment as assessed by physical examination and a stable health status. The laboratory values must be within the normal range of the assessing site or show abnormalities that are deemed not clinically significant as judged by the investigator. A stable health status is defined as the absence of a health event satisfying the definition of a serious adverse event.
3. Accessible vein for blood collection.
4. Subjects who are willing to comply with the requirements of the study protocol and scheduled visits. (e.g., completion of the subject diary, return for follow-up visits) and who are willing to make themselves available for the duration of the study, with access to a consistent means of telephone contact, which may be either at home or at the workplace, land line, or mobile, but NOT a pay phone or other multiple-user device (i.e. a common-use phone serving multiple rooms or apartments).
5. Ability to provide informed consent
6. Female subjects of non-child bearing potential due to surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or menopause. Post-menopausal subjects must have had at least 12 months of natural (spontaneous) amenorrhea.
7. Female subjects of childbearing potential may be enrolled in the study if they have negative urine pregnancy tests on the day of screening and day of antibiotic administration.
8. Willing to abstain from the use of probiotics or prebiotics for the duration of the study.

Exclusion Criteria:

1. Underlying chronic medical illness
2. History of Clostridium difficile diarrhea
3. History of Inflammatory Bowel disease or any other chronic gastrointestinal tract illness
4. Known drug allergy to amoxicillin-clavulanate, its components, or any other beta-lactam antibiotics.
5. Presence of acute infection in the preceding 7 days or presence of a temperature ≥ 38.0°C (oral or tympanic temperature assessment), or acute symptoms greater than of "mild" severity on the scheduled date of first dose
6. Any condition that, in the opinion of the investigator, would complicate or compromise the study or wellbeing of the subject.
7. Woman who is pregnant or breast feeding.
8. Evidence of substance abuse, or previous substance abuse including alcohol
9. Participation in a study involving administration of an investigational compound within the past three months, or planned participation during the duration of this study.
10. Receipt of antibiotics in the past 3 months.
11. Receipt of probiotics or prebiotics in the past 7 days.
12. Previous history of Augmentin-associated jaundice and/or hepatic dysfunction.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Operational taxonomic unit counts of bacterial species in the gut microbiota | 28 days
  Change from baseline in operational taxonomic unit counts of bacterial species in the gut microbiota of subjects who develop AAD compared to those who do not develop AAD after a 3 day course of oral Augmentin

SECONDARY OUTCOMES:
Diversity index of gut microbiome | 28 days
  Change from baseline in diversity index of gut microbiota of subjects who develop AAD compared to those who do not develop AAD after a 3 day course of oral Augmentin.

CONTACTS AND LOCATIONS:
Overall Officials: Shirin Kalimuddin, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No